CLINICAL TRIAL: NCT02980510
Title: Phase II Randomized Study Comparing FOLFIRINOX + Panitumumab Versus mFOLFOX6 + Panitumumab in Metastatic Colorectal Cancer Patients Selected by RAS and B-RAF Status From Circulating DNA Analysis
Brief Title: Comparison FOLFIRINOX Panitumumab vs mFOLFOX6 Panitumumab in RAS/B-RAF Wild-type Metastatic Colorectal Cancer Patients
Acronym: PANIRINOX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCGI 28 PANIRINOX; 2016-001490-33 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Oxaliplatin; Leucovorin; Irinotecan

STUDY DESIGN:
Intervention Model Description: National trial, multicenter, randomized, phase II assessing FOLFIRINOX + Panitumumab versus mFOLFOX6 + Panitumumab in metastatic colorectal cancer patients selected by RAS and B-RAF status from circulating DNA analysis.
Masking Description: The primary endpoint is the complete response rate where complete response is defined as complete disappearance of metastatic lesions after a maximum of 12 cycles of chemotherapy and tumor marker level normalization (CEA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A=Experimental group (Experimental): FOLFIRINOX + Panitumumab oxaliplatin 85 mg/m² IV infusion over 2 hours immediately followed by folinic acid 400 mg/m² given as a 2-hour intravenous (IV) infusion with the addition, after 30 minutes of irinotecan 150 mg/m² given as a 90-minute intravenous infusion through a Y-connector immediately followed by fluorouracil 400 mg/m² IV bolus then 5-fluoruracil (5-FU) 2400 mg/m² over 46 hours continuous infusion.
  Interventions: Drug: Panitumumab, oxaliplatin, folinic acid, 5-fluoruracil, irinotecan
- B=Control group (Active Comparator): mFOLFOX6 + Panitumumab mFOLFOX6 every 2 weeks: oxaliplatin 85 mg/m² IV infusion over 2 hours immediately followed by folinic acid 400 mg/m² IV infusion over 2 hours followed by fluorouracil 400 mg/m² IV bolus then 5-FU 2400 mg/m² over 46 hours continuous infusion.
  Interventions: Drug: Panitumumab, oxaliplatin, folinic acid, 5-fluoruracil

INTERVENTIONS:
Drug: Panitumumab, oxaliplatin, folinic acid, 5-fluoruracil
  Arms: B=Control group
Drug: Panitumumab, oxaliplatin, folinic acid, 5-fluoruracil, irinotecan
  Arms: A=Experimental group

SUMMARY:
National trial, multicenter, randomized, phase II assessing FOLFIRINOX + Panitumumab versus mFOLFOX6 + Panitumumab in metastatic colorectal cancer patients selected by RAS and B-RAF status from circulating DNA analysis.

Evaluation of complete response rate on treatment combining FOLFIRINOX and panitumumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: Evaluation of complete response rate on treatment combining FOLFIRINOX and panitumumab

SECONDARY OBJECTIVE(S):

* Overall Survival
* Progression free survival
* Secondary resection
* Early tumor shrinkage (ETS)
* Depth of response (DpR)
* Safety profile (NCI-CTCAE v4.03 classification)
* Diagnostic performance of ccfDNA analysis compared to the tumor-tissue analysis (current gold standard)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. ECOG PS between 0 and 1
3. Histologically confirmed adenocarcinoma of the colon or rectum
4. Untreated synchronous or metachronous metastatic disease deemed unresectable with curative intent
5. K-Ras (codons 12, 13, 59, 61, 117, 146), N-Ras (codons 12, 13, 59, 61) and B-Raf (codon 600) wild-type tumor status according to plasma analysis of circulating cell free DNA by Intplex technology
6. Measurable disease according to RECIST version 1.1
7. Adequate hematologic, hepatic and renal functions:

   * Absolute neutrophil count (ANC) ≥2 x 109/L
   * Haemoglobin ≥9 g/dL
   * Platelets (PTL) ≥100 x 109/L
   * AST/ALT ≤5 x ULN
   * Alkaline phosphatase ≤2.5 x ULN
   * Bilirubin ≤1.5 x ULN
   * Creatinine clearance ≥50 mL/min (Cockcroft and Gault formula)
8. Life expectancy of at least 3 months
9. Adequate contraception if applicable
10. Patient affiliated to a social security regimen
11. Patient information and signed written consent form
12. Uracilemia < 16 ng/ml

Exclusion Criteria:

1. History of other malignancy within the previous 5 years (except for appropriately treated in-situ cervix carcinoma and non-melanoma skin carcinoma)
2. Adjuvant treatment with oxaliplatin
3. Previous treatment for metastatic disease
4. Patients who received any chemo- and/or radiotherapy within 15 days from the date of blood sampling for the RAS and BRAF test
5. Brain metastases
6. Patients with a history of severe or life-threatening hypersensitivity to the active substances or to any of the excipients delivered in this study
7. Patient with history of pulmonary fibrosis or interstitial pneumonitis
8. Previous organ transplantation, HIV or other immunodeficiency syndromes
9. Concomitant medications/comorbidities that may prevent the patient from receiving study treatment as uncontrolled intercurrent illness (for instance: active infection, active inflammatory disorders, inflammatory bowel disease, intestinal obstruction, symptomatic congestive heart failure, uncontrolled hypertension…)
10. Persistent peripheral neuropathy >grade1 (NCI CT v4.03)
11. Ionic disorders as:

    * Kalemia ≤1 x LLN
    * Magnesemia <0.5mmol/L
    * Calcemia <2mmol/L
12. Patient with known dihydropyrimidine dehydrogenase deficiency
13. QT/QTc>450msec for men and >470msec for women
14. Patient with contraindication for trial drugs (investigators have to refer to SmPC drugs, see Appendix 7)
15. Concomitant intake of St. John's wort
16. Other concomitant cancer
17. Participation in another therapeutic trial
18. Pregnant woman or lactating woman
19. Patients with psychological, familial, sociological or geographical condition hampering compliance with the study protocol and follow-up schedule
20. Legal incapacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of complete response rate on treatment combining FOLFIRINOX and panitumumab. | 12 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Thibault MAZARD, Principal Investigator — ICM VAL D'AURELLE
Locations (6):
- France (6):
  - Institut Sainte Catherine, Avignon
  - Centre Léon Berard, Lyon
  - Chu Saint Eloi, Montpellier
  - ICM Val D'Aurelle, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - CHU Carémeau - Institut de Cancérologie du Gard, Nîmes

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Pisareva E, Mihalovicova L, Pastor B, Kudriavtsev A, Mirandola A, Mazard T, Badiou S, Maus U, Ostermann L, Weinmann-Menke J, Neuberger EWI, Simon P, Thierry AR. Neutrophil extracellular traps have auto-catabolic activity and produce mononucleosome-associated circulating DNA. Genome Med. 2022 Nov 28;14(1):135. doi: 10.1186/s13073-022-01125-8. PMID 36443816